CLINICAL TRIAL: NCT07368868
Title: Effect of Ultraprotective Ventilation After Veno-venous ECMO Initiation on Urine Output and Acute Kidney Injury (VENTURI) - a Retrospective Single Center Study
Brief Title: Effect of Initiation of Veno-venous ECMO on Urine Output and Acute Kidney Injury
Acronym: VENTURI
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2025-0269
Record Dates: First submitted 2026-01-20; First posted 2026-01-27 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: ARDS (Acute Respiratory Distress Syndrome); Acute Kidney Injury; ECMO
Keywords: ECMO; acute kidney injury; ARDS
MeSH Terms: conditions — Acute Lung Injury; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
With this study, the investigators want to find out whether the use of a "lung machine" (extracorporeal membrane oxygenation (ECMO)) togethet with giving the lungs "rest" (by minimizing ventilary support) in people with severe pneumonia has an effect on how well the kidneys work.

The investigators will use information that was already collected while patients were staying in the intensive care unit. Patients do not need to do anything additional or undergo any additional procedures for this study.

DETAILED DESCRIPTION:
Some people with severe pneumonia need to be admitted to the intensive care unit. In very serious cases, the lungs may work so poorly that breathing without help is no longer possible. These patients then receive support from a breathing machine (a ventilator). Sometimes even this support is not enough, and a special machine is needed to temporarily take over the function of the lungs. This machine is called a "lung machine" (also known as ECMO).

When a patient is connected to this lung machine, the patient's own lungs are exposed to as little pressure and stimulation as possible. This is called "lung rest" and gives the lungs time to heal.

In people who are very ill, such as those with severe pneumonia, other organs can also be affected. The kidneys, which are important for making urine and removing waste products from the body, may suddenly stop working as well as they should. This study will examine whether using the lung machine and lung rest affects how the kidneys work.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Admission to the Intensive Care Unit (ICU) of Ghent University Hospital
* Treatment with veno-venous extracorporeal membrane oxygenation (VV- ECMO)
* ICU admission between 1 January 2019 and 31 December 2023

Exclusion Criteria:

* Receipt of renal replacement therapy (RRT) prior to ICU admission
* Patients already receiving VV-ECMO at the time of admission to the ICU of Ghent University Hospital (i.e., patients referred from another hospital on VV-ECMO)
* Patients who received VV-ECMO immediately upon admission to the ICU of Ghent University Hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted on the ICU of Ghent Univesity Hospital with acute respiratory distress who received support by veno-venous ECMO between 1 January 2019 and 31 December 2023
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2025-12-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Difference in urine output (staged by KDIGO criteria) 6h before and after start veno-venous ECMO and ultraprotective ventilation | 6 hours
  The difference in urine output will be investigated before and after start of veno-venous ECMO together with the initiation of ultraprotective ventilation. To compare the difference in urine output a timeframe of 6 hours before ECMO wil be compared to a timeframe six hours after ECMO initiation. The 6 hour timeframe was choosen because this is the duration of the AKI KDIGO stage 1 urine output criterium.

SECONDARY OUTCOMES:
Difference in urine output (staged by KDIGO criteria) 12h before and after start veno-venous ECMO and ultraprotective ventilation. | 12 hours
  The difference in urine output will be investigated before and after start of veno-venous ECMO together with the initiation of ultraprotective ventilation. To compare the difference in urine output a timeframe of 12 hours before ECMO will be compared to a 12 hour timeframe after ECMO initiation. The 12 hour timeframe was choosen because this is the duration of the AKI KDIGO stage 2 urine output criterium.
Difference in urine output (staged by KDIGO criteria) 24h before and after start veno-venous ECMO and ultraprotective ventilation. | 24 hours
  The difference in urine output will be investigated before and after start of veno-venous ECMO together with the initiation of ultraprotective ventilation. To compare the difference in urine output a timeframe of 24 hours before ECMO will be compared to a 24 hour timeframe after ECMO initiation. The 24 hour timeframe was choosen because this is the duration of the AKI KDIGO stage 3 urine output criterium.
Difference in serum creatinine (staged by KDIGO criteria) 24h before and after start veno-venous ECMO and ultraprotective ventilation. | 24 hours
  The difference in serum creatinine will be investigated before and after start of veno-venous ECMO together with the initiation of ultraprotective ventilation. To compare the difference in serum creatinine a timeframe of 24 hours before ECMO will be compared to a 24 hour timeframe after ECMO initiation. Acute kidney injuri and it severity will be defined by the KDIGO definition and classification.

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent university hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No
Data of individuals will not be shared according to General Data Protection Regulation (GDPR)